CLINICAL TRIAL: NCT00003307
Title: A Phase II Open Label Trial of Amifostine Plus Fractionated Radiotherapy for Primary Prostate Adenocarcinoma (T1a-T3b, NoMo, PSA>10 ng/ml) to Estimate Acute Grade 2 Genitourinary and Gastrointestinal Toxicity
Brief Title: Radiation Therapy Plus Amifostine in Treating Patients With Primary Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James Oleson, M.D., Arizona Cancer Center at University of Arizona Health Science Center
Purpose: Treatment
Other Study IDs: CDR0000066254; P30CA023074 (NIH); UARIZ-HSC-9817; ALZA-98-005-ii; NCI-V98-1412
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2006-05

CONDITIONS: Prostate Cancer; Radiation Toxicity
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; radiation toxicity
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Amifostine; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Amifostine may protect normal cells from the side effects of radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy plus amifostine in treating patients with primary prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the incidence, grade, and time course of acute grade 2 or higher gastrointestinal and genitourinary toxicities in patients with primary prostate adenocarcinoma receiving amifostine plus fractionated radiotherapy. II. Determine the incidence and nature of toxicity associated with amifostine in these patients. III. Assess tumor response to this treatment in these patients. IV. Assess impotency rates following radiotherapy in these patients.

OUTLINE: This is an open label study. Patients receive fractionated radiotherapy five days per week for 7 weeks plus amifostine IV push over 5 minutes, 15 minutes before each radiation treatment. Patients are followed at 1 month after radiotherapy, and then every 3 months for at least 5 years.

PROJECTED ACCRUAL: There will be 25 patients accrued into this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed prostate adenocarcinoma Stage T1a-T3b N0 M0 disease PSA at least 10 ng/mL prior to treatment Must have a risk of seminal vesicle involvement between 10-25% No palpable or radiographic evidence of seminal vesicle involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Greater than 24 months Hematopoietic: Not specified Hepatic: SGOT and SGOT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No severe cerebrovascular disease or sustained hypotension not secondary to antihypotensive medication Other: No history of inflammatory bowel disease No history of malignancy other than nonmelanoma skin cancer No underlying medical or psychiatric illness that may impair ability to participate in study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the prostate area Surgery: No prior radical prostatectomy Other: No hypertensive medications if blood pressure less than 120/70

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1998-03; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Oleson, MD, PhD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States